CLINICAL TRIAL: NCT03518554
Title: A Phase 1, Multi-Center, Dose Escalation, Open-Label Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Preliminary Evidence of Antitumor Activity of JAB-3068 in Adult Patients With Advanced Solid Tumors
Brief Title: A First in Human, Dose Escalation Study of JAB-3068 （SHP2 Inhibitor） in Adult Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jacobio Pharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JAB-3068-01
Record Dates: First submitted 2018-04-06; First posted 2018-05-08 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Non-small Cell Lung Cancer; Head and Neck Cancer; Esophageal Cancer; Other Metastatic Solid Tumors
Keywords: JAB-3068; SHP2; advanced solid tumor; NSCLC; ESCC; HNSCC; PTPN11; EGFR; Colorectal cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Head and Neck Neoplasms; Esophageal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Noonan Syndrome; Colorectal Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JAB-3068 (SHP2 inhibitor) (Experimental): Daily oral administration of JAB-3068
  Interventions: Drug: JAB-3068

INTERVENTIONS:
Drug: JAB-3068 — JAB-3068 will be orally administered on a daily basis. Patients need to fast 2 hours before （6 hours for PK days) and 2 hours after each dosing.

SUMMARY:
This is a phase 1, multi-center, dose escalation, open-label study to evaluate the safety, tolerability, pharmacokinetics, and preliminary evidence of antitumor activity of JAB-3068 in adult patients with advanced solid.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent obtained prior to any study-related procedure being performed;
2. Age 18 years or older;
3. Patients with histologically or cytologically confirmed, advanced solid tumors which have progressed despite standard therapy or for whom no standard therapy exists;
4. Patients with life expectancy ≥3 months;
5. Patients must have at least one measurable lesion as defined by RECIST v1.1;
6. Eastern Cooperative Oncology Group performance score 0 or 1;
7. Patients who have sufficient baseline organ function.

Exclusion Criteria:

1. Patients with life-threatening autoimmune disease or with autoimmune disorder and who are on long-term steroid treatment;
2. History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO;
3. Known malignant central nervous system (CNS) disease other than neurologically stable, treated brain metastases;
4. Active infection including hepatitis B, hepatitis C and human immunodeficiency virus (HIV)
5. Patients who have any severe and/or uncontrolled medical conditions or other conditions that, in the opinion of the Investigator and Sponsor, could affect the patient's participation in the study
6. Patients who have impaired cardiac function or clinically significant cardiac diseases;
7. Use of anti-cancer treatment drug ≤21 days or 5 half-lives (whichever is shorter) prior to the first dose of JAB-3068;
8. Use of an investigational drug during the past 30 days or 5 half-lives (whichever is shorter) prior to the first dose of JAB-3068;
9. No other anti-cancer therapy (chemotherapy, immunotherapy, hormonal therapy radiotherapy (except for palliative local radiotherapy), biological therapy or other novel agent is to be permitted while the patient is receiving study medication.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-04-23 (Actual); Primary Completion 2022-02-03 (Actual); Study Completion 2022-02-03 (Actual)

PRIMARY OUTCOMES:
Number of participants with dose limiting toxicities | up to 28-day per cycle
  Incidence of dose limiting toxicities (DLTs) in the dose escalation phase. A DLT is defined as an adverse event or abnormal laboratory value assessed as unrelated to disease, disease progression, inter-current illness, or concomitant medications that occurs within the first treatment cycle with JAB-3068.

SECONDARY OUTCOMES:
Number of participants with adverse events | Approximately 2 years
  All patients participating in this study will be assessed for incidence and severity of adverse events (AEs) and serious AEs, including changes in laboratory values, vital signs, electrocardiograms, cardiac imaging and ophthalmological assessments
Area under the curve | Approximately 2 years
  Area under the plasma concentration time curve of JAB-3068
Cmax | Approximately 2 years
  Highest observed plasma concentration of JAB-3068
Tmax | Approximately 2 years
  Time of highest observed plasma concentration of JAB-3068
T1/2 | Approximately 2 years
  Half life of JAB-3068
Objective response rate | Approximately 2 years
  ORR is defined as the proportion of participants with complete response or partial response (CR+PR)
Duration of response | Approximately 2 years
  DOR is defined as the time from the participant's initial objective response (CR or PR) to study drug therapy, to disease progression or death due to any cause, whichever occurs first.

OTHER OUTCOMES:
pERK | Approximately 2 years
  On treatment versus baseline comparison of pharmacodynamic marker pERK (Phosphorylated form of Extracellular signal-regulated kinase) on newly obtained tumor biopsy samples by IHC.

CONTACTS AND LOCATIONS:
Overall Officials: Jacobio Pharmaceuticals, Study Director — Jacobio Pharmaceuticals Co., Ltd.
Locations (4):
- United States (4):
  - HealthONE Clinic Services Oncology-Hematology, Denver, Colorado
  - Florida Cancer Specialists, Sarasota, Florida
  - Sarah Cannon Research Institute, Nashville, Tennessee
  - The University of Texas M. D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided